CLINICAL TRIAL: NCT07251283
Title: Food Insecurity and Eating Behavior Among Adults Receiving Buprenorphine or Methadone Maintenance Treatment: Pilot Study 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Stacey C. Sigmon, Professor, PI, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003125
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Food Security
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-groups pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Education (NE) control condition (No Intervention): Nutritional Education (NE) participants received brief education, a list of FI-related resources in their community, and assistance with contacting those resources.
- Nutritional Eduction + Meal Delivery (NE+MD) experimental condition (Experimental): NE + Meal Delivery (NE+MD) participants received the same educational platform plus weekly meal deliveries using a commercial service that delivers premade, refrigerated meals directly to the participant's home.
  Interventions: Other: NE + Meal Delivery (NE+MD) intervention

INTERVENTIONS:
Other: NE + Meal Delivery (NE+MD) intervention — NE + Meal Delivery (NE+MD) participants received the same educational platform plus weekly meal deliveries using a commercial service that delivers premade, refrigerated meals directly to the participant's home.
  Arms: Nutritional Eduction + Meal Delivery (NE+MD) experimental condition

SUMMARY:
The goal of this study is to evaluate the effects of a novel, mail-based meal delivery intervention among individuals receiving MOUD on household food security status. The main question it aims to answer is:

* Will participants randomized to the NE+MD intervention will demonstrate greater reductions in USDA FSS scores from intake to Study Week 24 than NE participants?

Participants with OUD and FI will be randomly assigned to one of two 24-week experimental conditions: Nutritional Education alone (NE) or NE + Meal Delivery (NE+MD).

NE control participants will receive brief NE, a list of FI-related resources in their community, and assistance with contacting any resources of interest.

NE+MD participants will receive the same educational platform plus commercial weekly meal deliveries directly to the participant's home (6 meals per week per household member).

All participants will complete monthly follow-up assessments throughout the 24-week study measuring food security status, psychosocial functioning, and biometric measures of health. All participants will also complete monthly follow-up assessments for 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* receiving methadone or buprenorphine treatment for OUD
* meet criteria for current FI as measured by the 18-item US Household Food Security Survey (FSS; Economic Research Service, USDA, 2012)

Exclusion Criteria:

* Significant psychiatric or medical illness
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Household food insecurity | Monthly during the 6-month intervention period and monthly during the 6-month post-intervention follow-up monitoring period
  Household food insecurity as measured by the USDA Household Food Security Survey (FSS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No